CLINICAL TRIAL: NCT01133808
Title: Effectiveness of Rotavirus Immunization at the Community Level in Nicaragua
Brief Title: Effectiveness of Rotavirus Immunization in Nicaragua
Status: Completed | Type: Observational
Sponsor: Sylvia Becker-Dreps (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Thrasher Research Fund (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor-Investigator, Sylvia Becker-Dreps, Assistant Professor, Department of Family Medicine, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: 09-0371; K01TW008401-01 (NIH)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Diarrhea
Keywords: diarrhea; childhood; rotavirus; vaccine; Nicaragua
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples obtained from children who develop diarrhea during the course of the study. In addition, stool samples will also be collected from normal children to serve as controls in laboratory analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the investigators study is to compare the rates of childhood diarrhea at the community level before and after the rotavirus vaccination program in León, Nicaragua. From preliminary studies, the investigators anticipate about a 28% reduction in diarrhea following the vaccination program among children who received the vaccine, and a smaller reduction in diarrhea among children who did not receive the vaccine, due to the effects of "herd immunity". In addition, the investigators will collect stool samples from children who develop diarrhea in order determine the etiology of childhood diarrhea in the post-rotavirus immunization era.

ELIGIBILITY:
Inclusion Criteria:

* Age under 5 years, inclusion in health and demographic surveillance system (CIDS) in Leon, Nicaragua

Exclusion Criteria:

* Parents do not consent to child's participation

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under age 5 in Leon, Nicaragua
Sampling Method: Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Becker-Dreps, MD, Principal Investigator — University of North Carolina, Chapel Hill